CLINICAL TRIAL: NCT01669252
Title: A Phase II, Open-label, Single-arm, Exploratory Pharmacogenomic Study of Single Agent Eribulin (HALAVEN®) as Neoadjuvant Treatment for Operable Stage I-II HER2 Non-overexpressing Breast Cancer.
Brief Title: Pharmacogenomic Study of Neoadjuvant Eribulin for HER2 Non-overexpressing Breast Cancer
Acronym: NeoEribulin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SOLTI Breast Cancer Research Group (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOLTI-1007; 2012-000394-23 (EudraCT Number)
Record Dates: First submitted 2012-08-09; First posted 2012-08-20 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Eribulin; Neoadjuvant; PAM50; Triple-negative; Luminal A; Luminal B
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eribulin (Experimental): 1.23 mg/m2 eribulin ready to use solution (equivalent to 1.4 mg/m2 eribulin mesilate) IV on Days 1 and 8 of every 21-day cycle, for 4 cycles.
  Interventions: Drug: Eribulin

INTERVENTIONS:
Drug: Eribulin — 1.23 mg/m2 eribulin ready to use solution (equivalent to 1.4 mg/m2 eribulin mesilate) IV on Days 1 and 8 of every 21-day cycle, for 4 cycles.
  Other Names: Halaven(R)

SUMMARY:
This is a prospective, non-randomized, open-label, multicenter, single-arm exploratory pharmacogenomic study of single agent eribulin as neoadjuvant therapy in patients with operable Stage III HER2 non-overexpressing breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent, specifically highlighting the molecular characterization of tumor and genomic samples
* Age ≥18 years
* Histologically confirmed invasive breast carcinoma, with all of the following characteristics:

  * Primary tumor ≥2cm in largest diameter (cT1-3)
  * cN0-1
  * No evidence of distant metastasis (M0)
* Breast cancer (BC) eligible for primary surgery
* Available pre-treatment core (Tru-cut) biopsy or possibility of performing one
* HER2-negative BC (as per local assessment), defined as either of the following:

  * 0-1+ expression by IHC
  * 2+ expression by IHC and in situ hybridization (FISH/CISH) without HER2 gene amplification (<4 HER2 gene copies per nucleus, or a FISH ratio [HER2 gene copies to Cr17 signals] of <1.8)
  * Is situ hybridization (FISH/CISH) without HER2 gene amplification, independently of IHC
* Known hormone receptor (ER/PgR) status (as per local assessment) or the possibility of performing the tests
* Known percentage of hormone receptor (ER/PgR) and Ki67-positive tumor cells (as per local assessment), or possibility of performing the tests
* In the case of a multifocal tumor, the largest lesion must be ≥2 cm and designated the "target" lesion for all subsequent tumor evaluations and HER2-negative status must be documented in all the tumor foci
* ECOG performance status of 0 or 1
* Laboratory values as follows:

  * Absolute neutrophil count (ANC) ≥1.5 x 109/L
  * Platelets count ≥100 x 109/L
  * Hemoglobin ≥9 g/dL
  * Serum bilirubin ≤1.5 time the upper limit of normal (ULN)
  * Alanine aminotransferase and aspartate aminotransferase (AST) ≤2.5 x ULN
  * Alkaline phosphatase ≤2.5 x ULN
  * Serum creatinine ≤1.5 mg/dL or calculated creatinine clearance ≥60 mL/m
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Ability and willingness to comply with study visits, treatment, testing, and to comply with the protocol
* Availability of genomic DNA (via whole blood)

Exclusion Criteria:

* Any prior treatment for primary invasive BC
* Metastatic, locally advanced or inflammatory (i.e., Stage III-IV) BC
* Bilateral invasive BC
* Multicentric BC, defined as the presence of two or more foci of cancer in different quadrants of the same breast
* Pre-existing peripheral neuropathy of any grade
* Uncontrolled hypertension (systolic >150 mmHg and/or diastolic >100 mmHg)
* Clinically significant (i.e., active) cardiovascular disease
* Long QT syndrome
* Concomitant use of inhibitors of hepatic transport proteins such as organic anion-transporting proteins, P-glycoprotein, multidrug resistant proteins etc
* Major medical conditions that might affect study participation (e.g., uncontrolled seizure disorder, uncontrolled pulmonary, renal or hepatic dysfunction, or uncontrolled infection)
* Other primary malignant tumors within the previous 5 years, except for adequately controlled limited basal cell carcinoma of the skin or carcinoma in situ of the cervix
* Known human immunodeficiency virus(HIV) infection or other active or serious infection requiring IV antibiotics at randomization
* Pregnancy or breastfeeding women
* Women of childbearing potential(<2 years after the last menstruation) not using effective, non-hormonal means of contraception during the study and for a period of 6 months following the last administration of study drug
* Administration of any live virus vaccine within 8 weeks preceding study entry
* Use of any investigational agent within 30 days of administration of the first dose of study drug or concurrent treatment on another clinical study
* Requirement for radiation therapy concurrent with study anticancer treatment
* Known hypersensitivity to any of the study drugs or excipients
* Inability or unwillingness to abide by the study protocol or cooperate fully with the investigator or designee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2012-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Correlation of pre-treatment relative abundance of hundreds of mRNA transcripts from primary breast tumors with pCRB after neoadjuvant treatment with eribulin. | At the time of definitive surgery.
  pCRB , defined as the complete absence of invasive carcinoma in the breast on histological examination at the time of definitive surgery, according to the NSABP guidelines

SECONDARY OUTCOMES:
Rate of pCRB, defined as the complete absence of invasive carcinoma in the breast on histological examination at the time of definitive surgery, according to the NSABP guidelines. | At the time of definitive surgery
Rate of pCRBL, defined as the complete absence of invasive carcinoma in the breast and axillary lymph nodes on histological examination at the time of definitive surgery. | At the time of definitive surgery
Clinical and radiological ORR, defined by RECIST 1.1 | At the time of definitive surgery
Correlation of mRNA expression in breast tumors with clinical and radiological ORR at different time points during the neoadjuvant treatment with eribulin. | Up to 21 weeks
Rate of pCRB according to breast cancer subtype: Luminal A, Luminal B, Basal-like, HER2-enriched and Claudin-low. | At the time of definitive surgery
Rate of pCRB according to breast cancer subtype determined by immunohistochemistry (following the 2011 St. Gallen definitions): Luminal A, Luminal B, and TNBC. | At the time of definitive surgery
Proportion of patients able to have breast conservation surgery after being treated with eribulin as neoadjuvant therapy. | At the time of definitive surgery
The correlation between alternations in tubulin isotype expression and mutational status in pre-treatment samples with efficacy parameters, such as pCRB, ORR and BOR. | At the time of definitive surgery
The correlation between exome or genome sequencing data from pre-treatment samples with pCRB after neoadjuvant treatment with eribulin. | At the time of definitive surgery
Changes in gene expression and gene mutational status between the pre-treatment samples and samples after treatment. | At the time of definitive surgery
Number of participants with AEs and serious AEs (assessed by CTCAE v.4) | Up to 21 weeks
Percentage of patients who had neutropenia Grade 3-4 | Up to 21 weeks
Percentage of subjects with neuropathy | Up to 21 weeks
Incidence of dose reductions and/or dose delays due to treatment toxicity | Up to 71 days
Analysis of the expression of mRNA from breast tumors | At screening
Analysis of the expression of mRNA from breast tumors | At 21 days
Analysis of the expression of mRNA from breast tumors | At the time of definitive surgery
Correlation of mRNA expression in breast tumors after 21 days of neoadjuvant treatment and at surgery with pCRB. | At the time of definitive surgery
Sensitivity of the gene expression analysis of samples to predict clinical response to eribulin. | At screening
Sensitivity of the gene expression analysis of samples to predict clinical response to eribulin. | At 21 days
Sensitivity of the gene expression analysis of samples to predict clinical response to eribulin. | At time of definitive surgery
Specificity of the gene expression analysis of samples to predict clinical response to eribulin. | At screening
Specificity of the gene expression analysis of samples to predict clinical response to eribulin. | At 21 days
Specificity of the gene expression analysis of samples to predict clinical response to eribulin. | At time of definitive surgery

CONTACTS AND LOCATIONS:
Overall Officials: Javier Cortés, MD, Principal Investigator — Hospital Universitario Vall d´Hebron; Aleix Prat, MD, Principal Investigator — Vall d´Hebron Institut d´Oncologia
Locations (29):
- Institut Gustave Roussy, Villejuif, France
- Germany (4):
  - Brustzentrum im Krankenhaus Köln-Holweide Priv. Doz., Cologne
  - Klinikum des Landkreises Deggendorf Frauenklinik Mammazentrum, Deggendorf
  - Brustzentrum der Universität München, Munich
  - Klinikum Südstadt Rostock, Universitätsfrauenklinik und Poliklinik, Rostock
- Portugal (3):
  - Instituto Portugues de Oncologia de Coimbra Francisco Gentil, EPE, Coimbra
  - Hospital da Luz, Lisbon
  - Instituto Portugues de Oncologia de Porto Francisco Gentil, EPE, Porto
- Spain (21):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d´Hebron, Barcelona
  - Complejo Hospitalario de Castellón, Castellon
  - Complejo Hospitalario San Pedro de Alcántara, Cáceres
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Marina Salud de Denia, Denia
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro de Majadahonda, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitari Sant Joan de Reus, Reus
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital Virgen de la Macarena, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital de Torrevieja, Torrevieja
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Arnau de Vilanova de Valencia, Valencia
  - Hospital Universitario Lozano Blesa, Zaragoza

REFERENCES:
- [Background] Prat P, Llombart A, de la Peña L, Di Cosimo S, Oliveira M, Ortega V, Rubio I, Muñoz E, Harbeck N, Cortés J. NeoEribulin: A Phase II, non-randomized, open-label, single-arm, multicenter, exploratory pharmacogenomic study of single agent eribulin as neoadjuvant treatment for operable Stage I-II HER2 non-overexpressing breast cancer. Poster session presented at: 35th Annual San Antonio Breast Cancer Symposium (SABCS); 2012 December 4th-8th; San Antonio, Texas, United States.
- See also: SOLTI Breast Cancer Research Group — http://www.gruposolti.org